CLINICAL TRIAL: NCT06435884
Title: Long-Term Follow-up of Adult With Atrophic Scars Treated With TRTP-101 in Study CIC101-01
Brief Title: Long-Term Follow-up of Adult With Atorpphic Scars Treated With TRTP-101
Status: Recruiting | Type: Observational
Sponsor: CellinCells (Industry)
Responsible Party: Sponsor
Other Study IDs: CIC101-01-LT
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Atrophic Scar

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CIC101-01-LT is a long-term follow-up study of subjects treated with TRTP-101 and will evaluate the long-term safety and efficacy of TRTP-101.

DETAILED DESCRIPTION:
The long-term safety of TRTP-101 was evaluated by participants in the CIC101-01 clinical trial and followed up for 5 years for serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Received TRTP-101 in clinical trial CIC101-01
* Provided written informed consent to participate in this study

Exclusion Criteria:

* Judged to be unsuitable to participate in this long-term follow-up

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with Atropic Scars Treated with TRTP-101 in Sutdy CIC101-01
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Event | Up to 5 years
  SAE will be collected

SECONDARY OUTCOMES:
Mean percent change in atrophic scar volume | 6, 12, 18 and 24 months
  The depressed volume of atropic scar is measured at baseline in study CIC101-01
Patient's Satisfaction | 6, 12, 18 and 24 months
  Patient's Satisfaction with treatment scored by a 100-mm VAS(Visual Analogie Scale). On this scale, 0 indicates no satisfaction and 100 indicate extreme satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: JongHee Lee, MD, Principal Investigator — Department of Dermatology, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea